CLINICAL TRIAL: NCT05789147
Title: EffecTs of tRanscutaneous vAgus Nerve Stimulation in Heart Failure Patients With Moderately rEduced or preseRved Left Ventricular Function
Brief Title: Transcutaneous Vagus Nerve Stimulation in Heart Failure
Acronym: TRANSFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE 2182; RF-2016-02364803 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2023-02-28; First posted 2023-03-29 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Heart Failure With Midrange Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Randomized controlled study to evaluate the effects of 6-month tVNS (1 hour/day) in heart failure patients on autonomic biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tVNS (Active Comparator): Patients randomized to active treatment will be instructed to receive the stimulation at the tragus
  Interventions: Device: Active tVNS
- sham tVNS (Placebo Comparator): Patients randomized to active treatment will be instructed to receive the stimulation at the ear lobe
  Interventions: Device: Sham tVNS

INTERVENTIONS:
Device: Active tVNS — It is a non-invasive transcutaneous electrical stimulation of the auricular branch of the vagus nerve which innervates the skin of the human ear. These nerve fibers project directly to the solitary tract nucleus (NTS) in the brain stem (6).
  Arms: active tVNS
Device: Sham tVNS — Sham stimulation is obtained by placing the stimulation electrode at the level of the earlobe. The stimulation is therefore administered and perceived in an area not innervated by vagal fibers.
  Arms: sham tVNS

SUMMARY:
Several studies have shown that alterations in autonomic nervous system function are implicated in the onset and progression of numerous cardiovascular diseases. Direct stimulation of the vagus nerve by means of a sleeve placed around the vagus nerve represents one of the methodologies proposed in the field of neuromodulation. This study, which is proposed as a pilot study for further application of the method in subjects with cardiovascular disease aims to verify and consolidate evidence on cardiovascular autonomic effects in patients with heart failure. Vagal stimulation will be achieved noninvasively by applying an external stimulator to the auricular site.

DETAILED DESCRIPTION:
The autonomic nervous system (ANS), through the interaction between the sympathetic and vagal systems, plays a key role in modulating the cardiovascular system. Multiple experimental data and clinical studies have shown that alterations in the activity of the ANS - characterized by a predominant sympathetic modulation associated with reduced vagal modulation - are implicated in the onset and progression of numerous cardiovascular diseases. For example, both an increase in sympathetic activity and a reduction in vagal activity are associated with an increased risk of death after myocardial infarction and heart failure, and a further reduction in vagal activity has been shown to precede the phases of hemodynamic instability (1 -2).

Over the last few years, the modulation of the ANS through the implantation of devices has emerged as a new frontier for the treatment of heart failure (3). Although there is a wide interest in the scientific community for the potential represented by this therapeutic modality, nevertheless the different devices for neuromodulation therapy are implantable devices (whose application requires an invasive procedure) and therefore not free from risks and complications.

Direct stimulation of the vagus nerve by means of a sleeve positioned around the vagus nerve in its right or left cervical portion and controlled by a pacemaker, represents one of the methods proposed in the field of neuromodulation (4).

As for vagal stimulation, this can also be achieved non-invasively by applying an external stimulator in the ear (5). Transcutaneous nerve stimulation is a widely used procedure for the treatment of refractory epilepsy, while there is still limited experience evaluating its cardiovascular effects. Preliminary data in healthy volunteers have shown that: a) transcutaneous vagal stimulation, through the auricle, is able to activate the afferent vagal pathway up to the nucleus of the solitary tract (6), b) non-invasive stimulation of the vagus nerve is able to reduce sympathetic outflow (7). Recent clinical experience suggests its role also in the control of paroxysmal atrial fibrillation (8).

Therefore, non-invasive vagus nerve stimulation could be a promising therapeutic option in the cardiovascular field.

This study aims to evaluate the effects of long-term transcutaneous vagus nerve stimulation (tVNS) on autonomic parameters and other available physiological biomarkers that reflect long-term adjustment of autonomic neural regulation and to correlate the magnitude of the response to the baseline autonomic profile. A preliminary set of experiments will be conducted on healthy subjects to define the best tVNS protocol (in terms of frequency and site of stimulation) to induce acute changes in the autonomic profile.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients with moderately reduced or preserved ejection fraction
* Sinus rhythm
* New York Heart Association (NYHA) Class II-III

Exclusion Criteria:

* Patients with implanted cardiac device (ICD, CRT),
* Patients with recent (< 3 months) cardiac surgery,
* Patients with recent (< 3 months) myocardial infarction,
* Patients with recent (< 3 months) revascularization
* Patients with an indication for cardiac surgery within the next 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 6 months
  beats/min

SECONDARY OUTCOMES:
Baroreflex Sensitivity | 6 months
  ms/mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri IRCCS, Pavia, PV, Italy

REFERENCES:
- [Background] La Rovere MT, Bigger JT Jr, Marcus FI, Mortara A, Schwartz PJ. Baroreflex sensitivity and heart-rate variability in prediction of total cardiac mortality after myocardial infarction. ATRAMI (Autonomic Tone and Reflexes After Myocardial Infarction) Investigators. Lancet. 1998 Feb 14;351(9101):478-84. doi: 10.1016/s0140-6736(97)11144-8. PMID 9482439
- [Background] Mortara A, La Rovere MT, Pinna GD, Prpa A, Maestri R, Febo O, Pozzoli M, Opasich C, Tavazzi L. Arterial baroreflex modulation of heart rate in chronic heart failure: clinical and hemodynamic correlates and prognostic implications. Circulation. 1997 Nov 18;96(10):3450-8. doi: 10.1161/01.cir.96.10.3450. PMID 9396441
- [Background] Schwartz PJ, La Rovere MT, De Ferrari GM, Mann DL. Autonomic modulation for the management of patients with chronic heart failure. Circ Heart Fail. 2015 May;8(3):619-28. doi: 10.1161/CIRCHEARTFAILURE.114.001964. No abstract available. PMID 25991804
- [Background] Klein HU, Ferrari GM. Vagus nerve stimulation: A new approach to reduce heart failure. Cardiol J. 2010;17(6):638-44. PMID 21154273
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part II. Headache. 2016 Feb;56(2):259-66. doi: 10.1111/head.12650. Epub 2015 Sep 18. PMID 26381725
- [Background] Frangos E, Ellrich J, Komisaruk BR. Non-invasive Access to the Vagus Nerve Central Projections via Electrical Stimulation of the External Ear: fMRI Evidence in Humans. Brain Stimul. 2015 May-Jun;8(3):624-36. doi: 10.1016/j.brs.2014.11.018. Epub 2014 Dec 6. PMID 25573069
- [Background] Clancy JA, Mary DA, Witte KK, Greenwood JP, Deuchars SA, Deuchars J. Non-invasive vagus nerve stimulation in healthy humans reduces sympathetic nerve activity. Brain Stimul. 2014 Nov-Dec;7(6):871-7. doi: 10.1016/j.brs.2014.07.031. Epub 2014 Jul 16. PMID 25164906
- [Background] Stavrakis S, Humphrey MB, Scherlag BJ, Hu Y, Jackman WM, Nakagawa H, Lockwood D, Lazzara R, Po SS. Low-level transcutaneous electrical vagus nerve stimulation suppresses atrial fibrillation. J Am Coll Cardiol. 2015 Mar 10;65(9):867-75. doi: 10.1016/j.jacc.2014.12.026. PMID 25744003
- [Background] Maestri R, Pinna GD. POLYAN: a computer program for polyparametric analysis of cardio-respiratory variability signals. Comput Methods Programs Biomed. 1998 Apr;56(1):37-48. doi: 10.1016/s0169-2607(98)00004-2. PMID 9617526
- [Background] Pinna GD, Maestri R, Torunski A, Danilowicz-Szymanowicz L, Szwoch M, La Rovere MT, Raczak G. Heart rate variability measures: a fresh look at reliability. Clin Sci (Lond). 2007 Aug;113(3):131-40. doi: 10.1042/CS20070055. PMID 17381425
- [Background] Pinna GD, Maestri R, Raczak G, La Rovere MT. Measuring baroreflex sensitivity from the gain function between arterial pressure and heart period. Clin Sci (Lond). 2002 Jul;103(1):81-8. doi: 10.1042/cs1030081. PMID 12095408
- [Result] Maestri R, Pinna GD, Robbi E, Cogliati C, Bartoli A, Gambino G, Rengo G, Montano N, La Rovere MT. Impact of optimized transcutaneous auricular vagus nerve stimulation on cardiac autonomic profile in healthy subjects and heart failure patients. Physiol Meas. 2024 Jul 17;45(7). doi: 10.1088/1361-6579/ad5ef6. PMID 39016202